CLINICAL TRIAL: NCT04391790
Title: Randomized Controlled Trial With a MOdified Urinary Conduit to Lower Strictures After radIcal Cystectomy - MOSAIC
Brief Title: MOdified Urinary Conduit to Lower Strictures After radIcal Cystectomy
Acronym: MOSAIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jørgen Bjerggaard Jensen (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, Consultant, MD, DMSc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOSAIC; DaBlaCa-16 (Other: Danish Bladder Cancer Group)
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Bladder Cancer
Keywords: ureteral strictures; urinary diversion
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystectomy

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Study subject will cohere to current national guidlines with a cystectomy and standard urinary conduit ad modum Bricker
  Interventions: Procedure: Cystectomy and standard urinary conduit ad modum Bricker
- Intervention (Experimental): Subject in the interventional arm, will be treated with a cystectomy and modified retrosigmoid conduit
  Interventions: Procedure: Cystectomy and modified urinary conduit

INTERVENTIONS:
Procedure: Cystectomy and modified urinary conduit — The modified retrosigmoid conduit is extended aorund 5 cm, so the left ureter does not have to cross under the mesentery wheras the presumed more robust ileal segment does.
  Other Names: Retrosigmoid conduit
  Arms: Intervention
Procedure: Cystectomy and standard urinary conduit ad modum Bricker — The conduit is constructed using approximately 15 cm of terminal ileum and placed in the right side of the abdomen. In order for the left ureter to reach the conduit, it is mobilized behind the sigmoideum to the conduit.
  Other Names: Conventional ileal conduit
  Arms: Control

SUMMARY:
Cystectomy is the chosen treatment of bladder cancer in 400 cases every year in DK. In replacement of the removed bladder, a urinary diversion is constructed using 15cm of terminal ilium (Ad Modum Bricker).

Ureteral strictures are diagnosed in 15% of the cystectomized patients, and these patients are at increased risk of infections, loss of renal function and repeated interventions. The left ureter is diagnosed with 70% of all strictures, presumably due to the construction of the urinary diversion.

A modified urinary diversion have been tested in two small studies. The modified diversion is prolonged with 5cm compared to the conventional urinary diversion. The prolongation permits the urinary diversion to reach both the left and the right side of the abdomen, resulting in greater resection of non-viably distal ureter and less mobilization of the left ureter, lowering the rates of strictures.

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer with the indication for robot assisted radical cystectomy
* Ileal conduit ad modum Bricker as planned urinary diversion
* Ability to understand the participant information orally and in writing
* Signed consent form

Exclusion Criteria:

* Previous abdominal or pelvic radiotherapy
* Previous major abdominal surgery involving resection of bowel or construction of an enteric stoma
* Urostomy planned on the left side of the abdomen
* Single kidney
* Complete ureteral duplication (either uni- or bilaterally), known at time of inclusion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Strictures | Within 2 years after cystectomy
  Number of participants with benign strictures in the left ureter

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Department of Urology, Aalborg University Hospital, Aalborg
  - Department of Urology, Aarhus University Hospital, Aarhus
  - Department of Urology, Rigshospitalet, Copenhagen
  - Department of Urology, Herlev and Gentofte Hospital, Herlev
  - Department of Urology, Odense University Hospital, Odense